CLINICAL TRIAL: NCT01022736
Title: Preemptive Gabapentin Administration and Perioperative Plasma Concentrations With Cardiac Bypass
Brief Title: Plasma Gabapentin Concentration During and Following Cardiac Bypass
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Dr. Joel Parlow, Queen's University and Kingston General Hospital, Department of Anesthesiology & Perioperative Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANAE-128-06
Record Dates: First submitted 2009-11-27; First posted 2009-12-01 (Estimated); Last update posted 2009-12-08 (Estimated); Status verified 2009-12

CONDITIONS: Cardiopulmonary Bypass
Keywords: gabapentin; pharmacokinetics; visual analogue pain scale; cardiopulmonary bypass
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gabapentin (Experimental): patients scheduled for cardiac bypass surgery will be administered gabapentin (600mg, orally). Blood will be drawn and plasma gabapentin levels determined 1 hour before surgery, 10 minutes into surgery, 10 minutes before separation from bypass, 30 minutes following bypass, and then before and 2 hours after each dose of gabapentin.
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — Subjects will be administered gabapentin (600 mg, orally) 1 hour prior to cardiac bypass surgery, 1 hour following extubation, then every 8 hours for a total of 4 doses.
  Other Names: neurontin

SUMMARY:
This open label investigation is to determine whether cardiopulmonary bypass affects plasma gabapentin concentration after preoperative administration in the setting of cardiac bypass surgery. Following signed informed consent, 16 patients scheduled for cardiac bypass surgery will be given gabapentin (600mg, oral) 1 hour prior to surgery, 1 hour following extubation and then every 8 hours for a total of 4 doses. Plasma gabapentin levels will be measured prior to induction, prior to bypass, 10 min into the bypass procedure, 10 minutes before separation from bypass, 30 minutes following bypass and then before and 2 hours following each of the next 3 doses of gabapentin. Pain scores, sedation scores, side effects and morphine equivalents will be documented for one day following surgery.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for cardiac bypass surgery involving median sternotomy and CPB
* signed informed consent

Exclusion Criteria:

* history of chronic pain
* regular opioid consumption
* regular anticonvulsant consumption
* regular gabapentin or pregabalin use
* recent congestive heart failure
* ejection fraction <35%
* chronic pulmonary disease
* liver disease
* renal insufficiency (preoperative creatinine > 140umol/L
* history of adverse reaction to acetaminophen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-05; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
plasma concentrations of gabapentin | 1 hour before surgery, 10 min following initiation of bypass, 10 min before separation from bypass, 30 min following bypass, and then before and 2 hours following each of the next 3 doses of gabapentin

CONTACTS AND LOCATIONS:
Overall Officials: Joel Parlow, MD, Principal Investigator — Queen's University and Kingston General Hospital
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Parlow J, Gilron I, Milne B, Dumerton-Shore D, Orr E, Phelan R. Cardiopulmonary bypass does not affect plasma concentration of preoperatively administered gabapentin. Can J Anaesth. 2010 Apr;57(4):337-42. doi: 10.1007/s12630-010-9269-5. Epub 2010 Jan 29. PMID 20112079